CLINICAL TRIAL: NCT04280835
Title: The Effect of Group Psychoeducation That Focused on Social Skills Development Applied to Patients Who Diagnosed With Schizophrenia on Treatment Compliance, Quality of Life and Well-being
Brief Title: Psychoeducation in Patients Who Diagnosed With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Merve Kızılırmak Tatu, Principal Investigator, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKTatu
Record Dates: First submitted 2020-02-17; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Quality of Life; Well-Being; Compliance, Treatment
Keywords: schizophrenia; psychoeducation; compliance to treatment; quality of life; well-being
MeSH Terms: conditions — Patient Compliance; Schizophrenia

STUDY DESIGN:
Intervention Model Description: The research was using quasi-experimental research methods. The experimental group was composed of patients with schizophrenia registered at Community Mental Health Center and the control group was composed of outpatients diagnosed with schizophrenia who applied to Psychiatric Polyclinic.The patients met the inclusion criteria of the study and volunteered to participate in the study.The study was completed with 42 patients (n=21for the intervention group; n=21 patients for the control group).Psychoeducation program were applied to intervention group. No intervention was performed on the patients in the control group.To the experimental and control group, at screening (pre-test), eight weeks after screening (post-intervention/post-test), three months after the post tests (follow-up) was applied.The mesurements were taken simultaneously in the intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Psychoeducation that Focused on Social Skill Development (Experimental): The Psychoeducation program that focused on social skill development, consists of 8 sessions, one day a week, each lasting an average of 60 Minutes. Psychoeducation was conducted in three groups and each of them consisted of eight patients.
  Interventions: Behavioral: Group Psychoeducation that Focused on Social Skill Development
- Control Group (No Intervention): No intervention was performed on the patients in the control group, and routine follow-up (arranging treatment by the doctor, answering the patient's and family's questions about treatment) continued in the polyclinic.

INTERVENTIONS:
Behavioral: Group Psychoeducation that Focused on Social Skill Development — Psychoeducation Program consists of; Preparatory Session, Recognition of Schizophrenia, Evaluating the Treatment of Schizophrenia, Stress and Coping with Stress, Improving Communication Skills, Improving Problem-solving Skills, Improving Interpersonal relationships and social activities and Evaluating Session.The sessions were held in the form of PowerPoint presentations. In the psychoeducation program, lecture, question-answer, homework, sharing experiences, group discussion, repetition, video presentation, summarization, reinforcer, and role-playing techniques were used. The day before each session, patients were phoned and reminded of the time of the session. At the end of each session, the content of the subject is given as hard copy and cookies, tea and coffee were served.
  Arms: Group Psychoeducation that Focused on Social Skill Development

SUMMARY:
People with schizophrenia are faced with social problems such as repeated hospitalizations, stigma with lack of social skills, unemployment, lack of necessary and adequate health care and education due to lack of adequate care in the community they live in. It is known that psychoeducation practices aimed at developing social skills in schizophrenia give patients new skills and these skills continue for many years. This study aimed to determine the effect of group psychoeducation that focused on social skill development on treatment adaptation, quality of life and well-being in schizophrenia patients and the interaction between these variables over time.

DETAILED DESCRIPTION:
The aim is to determine the effect of group psychoeducation that focused on social skill development on treatment adaptation, quality of life and well-being in schizophrenia patients and the interaction between these variables over time.

The study was conducted with 42 schizophrenia patients (n=21 intervention group; n=21 control group) using a quasi-experimental research design. Patients were evaluated using a pre-test, post-test, monitoring test, "Medication Adherence Rating Scale (MARS)", "Quality of Life Scale for Schizophrenia (QLSS)" and "Flourishing Scale" (FS). The measurements were taken 3 times: pre test, post-test and 3-months post-test.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering
* Being 18 and over being literate
* Having been diagnosed with schizophrenia for at least three months
* Taking oral antipsychotics
* Being in remission.

Exclusion Criteria:

* Being in an acute period of exacerbation
* Actively using alcohol or psychoactive substances
* Having mental retardation or dementia
* Having another psychiatric illness that makes it impossible to cooperate.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life Scale for Schizophrenia (QLSS) | Change from baseline to 8 weeks (also assessed at 20 weeks post-baseline)
  It evaluates the quality of life of schizophrenic patients receiving maintenance treatment. QLSS provides information about ongoing symptoms and functionality. It is a 7-degree Likert type scale applied in a semi-structured interview format. It consists of a total of four sub-dimensions and 21 questions in the form of interpersonal relationships, professional role, psychic findings and daily item use-activities. The total score of all subscales gives the total score (0-126) of quality of life.
Medication Adherence Rating Scale (MARS) | Change from baseline to 8 weeks (also assessed at 20 weeks post-baseline)
  The scale assesses the patient's compliance behaviors and attitude to treatment. The scale consists of 10 questions to answer in the form of Yes/No (between 1-7 were poor in compliance with treatment and those with scores between 8-10 were high).
Flourishing Scale (FS) | Change from baseline to 8 weeks (also assessed at 20 weeks post-baseline)
  It is a self-assessment scale measures an individual's level of well-being. It consists of eight items and each item is scored 1-7 points. The total score range from 8-56 points. The more the score from the scale increases the more the well-being increases.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Kızılırmak Tatu, PhD, Principal Investigator — Gazi University Health Science Faculty, Ankara, Turkey.
Locations (1):
- Merve Kızılırmak Tatu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Other researchers will be able to read detailed information such as the research method and results when the research is published. The "Research Protocol" will be available on the this PRS page.